CLINICAL TRIAL: NCT00437320
Title: Comparison of Metvix PDT With Its Vehicle in the Treatment of Photoaged Skin
Brief Title: Comparison of Metvix Photodynamic Therapy (PDT) With Its Vehicle in the Treatment of Photoaged Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD.03.SPR.29057; 2006-004237-15 (EudraCT Number)
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-12

CONDITIONS: Photoaged Skin
Keywords: PDT; Photoaging; Galderma
MeSH Terms: interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metvix Cream 160 mg/g +Metvix Vehicle Cream (1 Hour Group) (Experimental): Participants were topically treated with 160 milligrams per gram (mg/g) Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 1 hour at Baseline, Weeks 4 and 8. The target area was then exposed to red light [using a large-field light emitting diode (LED) light source: Aktilite 128 lamp] during 7 to 10 minutes to deliver a total dose of 37 Joules per centimeter square J/cm^2. The total study duration was 20 weeks.
  Interventions: Drug: Metvix Cream 160 mg/g; Drug: Metvix Vehicle Group
- Metvix Cream 160 mg/g +Metvix Vehicle Cream (2 Hour Group) (Experimental): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 2 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
  Interventions: Drug: Metvix Cream 160 mg/g; Drug: Metvix Vehicle Group
- Metvix Cream 160 mg/g +Metvix Vehicle Cream (3 Hour Group) (Experimental): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
  Interventions: Drug: Metvix Cream 160 mg/g; Drug: Metvix Vehicle Group

INTERVENTIONS:
Drug: Metvix Cream 160 mg/g — Participants were treated with topical administration of Metvix cream.
  Other Names: methyl aminolevulinate
Drug: Metvix Vehicle Group — Participants were treated with topical administration of Metvix Vehicle cream.

SUMMARY:
Skin photoaging or skin photodamage were terms used to describe the change in the structure, function and appearance of skin caused by prolonged and repeated exposure to sunlight or other ultraviolet light sources.

The visible effects of skin photodamage were fine lines, skin sagging, skin roughness, liver spots and also the appearance of red patches made up of thin red vessels (called telangiectasia).

More and more people were presenting to doctors with concerns about skin photodamage and the demand for corrective procedures was increasing.

Metvix photodynamic therapy (Metvix PDT) is a procedure currently marketed in several countries in Europe (including the United Kingdom [UK] and Spain) and in Australia, for the treatment of benign forms of skin cancer (example, actinic keratosis).

The aim of the study was to assess whether Metvix PDT would be effective in correcting the effects related to photodamage and whether it would be well tolerated.

DETAILED DESCRIPTION:
Different application times of the study treatment were being investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants older than 30 years of age.
* Participants with a photodamage grade of at least 4 on the Griffiths photonumeric scale (symmetrical photodamage on the two target areas)
* Participants with mottled hyper-pigmentation on the face
* Participants willing and capable of cooperating to the extent and degree required by the protocol
* Participants must read the Patient Information Sheet and read and sign the Informed Consent form prior to any study related procedures.

Exclusion Criteria:

* Participants who were at risk in terms of precautions, warnings, and contra-indication in the package insert for Metvix
* Participants with suspected porphyria
* Participants with specific wash-out period for interfering treatments
* Participants requiring concurrent treatment that would interfere with study objectives and/or evaluations

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04-18 (Actual); Primary Completion 2008-09-01 (Actual); Study Completion 2008-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CEM Griffiths, Principal Investigator — Professor
Locations (3):
- Policlinico Ruber, Madrid, Spain
- United Kingdom (2):
  - Whittington Hospital, London
  - University of Manchester-Hope Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
The study protocol was submitted to and approved by the local Ethics Committees prior to study initiation, and by the regulatory authorities. The study was followed-up closely by the Sponsor or representatives according to the Declaration of Helsinki (1964) and its Tokyo 9(175), Venice (1983), Hong-Kong (1989), Somerset West (1996), and Edinburgh (2000) amendments, the ICH Good Clinical Practice (GCP) principles, Standard Operating Procedures (SOPs) and local regulatory requirements.

REFERENCES:
- See also: Related Info — http://www.metvix.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers in the United Kingdom and Spain from 18 April 2007 to 1 September 2008.
Pre-assignment Details: A total of 32 participants were enrolled in the study and randomized in three different groups (1 hour group, 2 hour group, and 3 hour group).
Units Other Than Participants: Half face
Groups:
- Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group): Participants were topically treated with 160 milligrams per gram (mg/g) Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 1 hour at Baseline, Weeks 4 and 8. The target area was then exposed to red light [using a large-field light emitting diode (LED) light source: Aktilite 128 lamp] during 7 to 10 minutes to deliver a total dose of 37 Joules per centimeter square J/cm^2. The total study duration was 20 weeks.
- Metvix Cream 160 mg/g+Metvix Vehicle Cream (2 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 2 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Cream 160 mg/g+Metvix Vehicle Cream (3 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
Period: Overall Study
Arm/Group | Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g+Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g+Metvix Vehicle Cream (3 Hour Group)
Started | 11; 11 Half face | 9; 9 Half face | 12; 12 Half face
Metvix Cream (1 Hour) | 11; 11 Half face | 0; 0 Half face | 0; 0 Half face
Metvix Vehicle Cream (1 Hour) | 11; 11 Half face | 0; 0 Half face | 0; 0 Half face
Metvix Cream (2 Hour) | 0; 0 Half face | 9; 9 Half face | 0; 0 Half face
Metvix Vehicle Cream (2 Hour) | 0; 0 Half face | 9; 9 Half face | 0; 0 Half face
Metvix Cream (3 Hour) | 0; 0 Half face | 0; 0 Half face | 12; 12 Half face
Metvix Vehicle Cream (3 Hour) | 0; 0 Half face | 0; 0 Half face | 12; 12 Half face
Completed | 9; 9 Half face | 8; 8 Half face | 8; 8 Half face
Not Completed | 2; 2 Half face | 1; 1 Half face | 4; 4 Half face
Not completed — Participant request | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled and randomized participants.
Groups:
- Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 1 hour at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Total: Total of all reporting groups
Arm/Group | Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g+Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g+Metvix Vehicle Cream (3 Hour Group) | Total
Number analyzed (Participants) | 11 | 9 | 12 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (7.3) | 57.0 (10.4) | 58.4 (9.3) | 59.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 10 | 27
  Male | 2 | 1 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 9 | 12 | 32
Phototype [Count of Participants; unit: Participants] — Skin phototype was used to describe a person's skin type. It ranges from skin phototype I to III. Where, skin phototype I = pale white skin, always burns easily, never tans; skin phototype II = fair skin, always burns easily, tans minimally and with difficulty; skin phototype III = darker white skin, burns minimally, tans gradually and uniformly.
  Participants
    Phototype I | 3 | 1 | 1 | 5
    Phototype II | 1 | 4 | 3 | 8
    Phototype III | 7 | 4 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severity of Photodamage
Description: Severity of cutaneous photodamage in participants were assessed using Griffiths photo numeric scale. The severity scores of photodamage on the scale ranged from 0 (minimum) to 8 (maximum), that is, no damage (0), mild damage (1-3), moderate damage (4-6), and severe damage (7-8) where the highest score indicated worst outcome.
Time Frame: At Week 20
Population: ITT population included all enrolled and randomized participants. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. As per planned analysis data was separately analyzed and collected for both Metvix cream and Metvix vehicle cream based on 1, 2 and 3 hours group."
Measure: Count of Participants; unit: Participants
Groups:
- Metvix Cream 160 mg/g (1 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face for 1 hour at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Vehicle Cream (1 Hour Group): Participants were topically treated with Metvix vehicle cream on the other half-face for 1 hour at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Cream 160 mg/g (2 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face for 2 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Vehicle Cream (2 Hour Group): Participants were topically treated with Metvix vehicle cream on the other half-face for 2 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Cream 160 mg/g (3 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Vehicle Cream (3 Hour Group): Participants were topically treated with Metvix vehicle cream on the other half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9
Participants
  No - Mild damage | 0 | 0 | 1 | 0 | 0 | 0
  Mild damage | 1 | 0 | 0 | 1 | 1 | 0
  Mild - Moderate damage | 0 | 0 | 1 | 1 | 0 | 1
  Moderate damage | 3 | 1 | 1 | 0 | 4 | 2
  Moderate - Moderate/ severe damage | 0 | 2 | 2 | 3 | 1 | 4
  Moderate/ severe damage | 2 | 3 | 1 | 1 | 3 | 2
  Moderate/ severe - Severe damage | 1 | 1 | 1 | 1 | 0 | 0
  Severe damage | 2 | 2 | 1 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Severity of Mottled Hyper-Pigmentation
Description: The evaluation of the severity of facial mottled hyperpigmentation were done using five-point scale. The score on the five-point scale ranged from 0 (minimum) to 4 (maximum), that is, 0 = none (no areas of mottled, irregular pigmentation), 1 = minimal (few, small lightly pigmented, discrete macules), 2 = mild (multiple, small lightly pigmented macules), 3 = moderate (widespread areas of mottled, moderately dark macules), 4 = severe (Widespread, multiple areas of dark macules/hyperpigmentation with uneven skin tone). The higher score indicated the worse outcome.
Time Frame: At Week 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Metvix Cream 160 mg/g (3 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9
Participants
  None | 1 | 0 | 0 | 0 | 1 | 0
  Minimal | 3 | 3 | 3 | 2 | 5 | 6
  Mild | 3 | 3 | 1 | 3 | 2 | 0
  Moderate | 2 | 2 | 4 | 3 | 1 | 3
  Severe | 0 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Severity of Fine Lines
Description: The evaluation of the severity of facial fine lines were done using the five-point scale ranging from 0 to 4, that is, 0 = none- (lines disappear with stretching), 1 = minimal (few lines which do not completely disappear with stretching), 2 = mild (few lines which only diminish with stretching), 3 = moderate (widespread areas of lines which change minimally with stretching), 4 = severe- (widespread areas of lines which do not change at all with stretching), where the higher score indicated the worse outcome.
Time Frame: At Week 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9
Participants
  Moderate | 3 | 7 | 2 | 3 | 4 | 4
  Severe | 1 | 0 | 0 | 1 | 0 | 1
  Mild | 2 | 2 | 4 | 3 | 2 | 1
  Minimal | 3 | 0 | 1 | 1 | 3 | 3
  None | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Severity of Telangiectasia
Description: The severity of telangiectasia by using the scale ranging from 0 (minimum) to 3 (maximum), that is, 0 = absent (no telangiectasia), 1 = mild (slight telangiectasia characterized by appearance of a few fine, small red vessels [0.2 millimeters [mm] or less in diameter); telangiectasia covers less than 10 percent (%) of the target area, 2 = moderate (pronounced telangiectasia characterized by appearance of several fine vessels and/or few large vessels [0.2 mm or greater in diameter]; telangiectasia covers between 10 to 30% of the target area), 3 = severe (severe telangiectasia characterized by the appearance of many fine vessels and/or large vessels; telangiectasia covers greater than 30% of the target area), where the higher score indicated the worse outcome.
Time Frame: At Week 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9
Participants
  Absent | 0 | 0 | 2 | 1 | 1 | 0
  Mild | 5 | 3 | 3 | 4 | 5 | 5
  Moderate | 4 | 6 | 3 | 2 | 3 | 4
  Severe | 0 | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Severity of Skin Roughness
Description: The evaluation of the severity of skin roughness were done by using the five-point scale ranging from 0 to 4,that is, 0 = none ( very smooth, no patches of roughness), 1 = minimal (smooth with only a few patches of roughness), 2 = mild (mostly smooth with scattered patches of roughness), 3 = moderate (slightly rough with diffuse patches of roughness), 4 = severe (rough with diffuse areas of roughness, some scales may be visible), where the higher score indicated the worse outcome.
Time Frame: At Week 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9 | 9
Participants
  None | 1 | 1 | 3 | 2 | 4 | 4
  Minimal | 5 | 2 | 1 | 1 | 2 | 0
  Mild | 2 | 2 | 4 | 4 | 2 | 3
  Moderate | 0 | 3 | 0 | 1 | 1 | 1
  Severe | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Participants With Severity of Skin Laxity
Description: The evaluation of the severity of skin laxity were done by using the scale ranging from 0 to 3 that is, 0 = none (no skin laxity), 1 = mild (mild skin sagging), 2 = moderate (moderate skin sagging), 3 = severe (severe skin sagging), where the higher score indicated the worse outcome.
Time Frame: At Week 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Metvix Vehicle Cream (3 Hour Group): Participants were topically treated with 160 mg/g Metvix vehicle cream on the other half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9
Participants
  None | 0 | 0 | 1 | 0 | 0 | 0
  Mild | 6 | 4 | 5 | 4 | 5 | 5
  Moderate | 2 | 4 | 1 | 2 | 4 | 3
  Severe | 1 | 1 | 1 | 2 | 0 | 1

7. Primary Outcome: Number of Participants With Tolerability Assessment of Erythema
Description: Erythema was defined as an abnormal redness of the skin and was measured on the scale score ranging from 0 (minimum) to 3 (maximum) that is, 0 = none (no erythema),1 = mild (slight pinkness present), 2 = moderate (definite redness, easily recognized), and 3 = severe (intense redness), where the higher score indicated the worse outcome.
Time Frame: At Week 20
Population: Safety population included all enrolled and randomized participants. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. As per planned analysis data was separately analyzed and collected for both Metvix cream and Metvix vehicle cream based on 1, 2 and 3 hours."
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 11 | 11
Participants
  None | 5 | 8 | 0 | 5 | 0 | 9
  Mild | 3 | 1 | 5 | 2 | 7 | 1
  Moderate | 1 | 0 | 4 | 2 | 3 | 1
  Severe | 0 | 0 | 0 | 0 | 1 | 0

8. Primary Outcome: Number of Participants With Tolerability Assessment of Edema
Description: Abnormal tenseness of the skin was measured on a scale ranging from 0 to 3. 0 (none) no edema, 1 (mild) slight tenseness of skin without firmness, 2 (moderate) moderate tenseness of the skin with slight firmness, 3 (severe) severe tenseness of the skin with resistance to distortion. The higher score means the worse outcome.
Time Frame: At Week 20
Population: Safety population included all enrolled and randomized participants. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. As per planned analysis data was separately analyzed and collected for both Metvix cream and Metvix vehicle cream based on 1, 2 and 3 hours group."
Measure: Count of Participants; unit: Participants
Groups:
- Metvix Vehicle Cream (2 Hour Group): Participants were topically treated with Metvix vehicle cream on the other half-face for 2 hours at Baseline, Week 20. The target area was then exposed to Aktilite 128 lamp for 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 11 | 11
Participants
  None | 5 | 8 | 5 | 7 | 4 | 10
  Mild | 3 | 1 | 2 | 2 | 6 | 0
  Moderate | 0 | 0 | 2 | 0 | 1 | 1
  Severe | 1 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Tolerability Assessment of Oozing/Crusting
Description: Oozing/crusting was a continuing process of exudation of fluid from the lesions/formation of scab-like material on the surface of lesions resulting from dried serum. Oozing/crusting was assessed on a scale ranging from 0-3. 0 (none) no oozing/crusting, 1 (mild) faint sign of oozing and/or weeping; slight crusting on a few of the lesions, 2 (moderate) definite oozing, but not extensive (a few lesions/areas); definite crusting on several of the lesions, 3 (severe) marked oozing/weeping; heavy crusting on the majority of the lesions. The higher score indicated the worse outcome.
Time Frame: At Week 20
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Metvix Vehicle Cream (2 Hour Group): Participants were topically treated Metvix vehicle cream on the other half-face for 2 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Cream160 mg/g (3 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix Vehicle Cream (3 Hour Group): Participants were topically treated Metvix vehicle cream on the other half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 11 | 11
Participants
  None | 8 | 9 | 7 | 8 | 6 | 10
  Mild | 1 | 0 | 2 | 1 | 2 | 1
  Moderate | 0 | 0 | 0 | 0 | 3 | 0

10. Primary Outcome: Participant's Skin Discomfort Score Using Visual Analogue Scale (VAS)
Description: Participant skin discomfort was evaluated on a scale of 0 to 10. 0 ("no skin discomfort") to 10 ("worst possible skin discomfort") evaluation of skin discomfort (including pain and itching) on each half-face was analyzed using a VAS. The higher score indicated the worse outcome.
Time Frame: At Week 4
Population: Safety population included all enrolled and randomized participants. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable for this OM at given timepoint. As per planned analysis data was separately analyzed and collected for both Metvix cream and Metvix vehicle cream based on 1, 2 and 3 hours group."
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 10 | 10
score on a scale | 3.0 (3.0) | 0 (0) | 4.6 (2.9) | 0.3 (0.7) | 6.3 (2.9) | 0.3 (0.4)

11. Primary Outcome: Participant's Skin Discomfort Score Using Visual Analogue Scale (VAS)
Description: as for outcome 10
Time Frame: At Week 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 10 | 10
score on a scale | 3.0 (2.9) | 0.0 (0.1) | 4.9 (2.6) | 0.0 (0.0) | 6.4 (2.3) | 0.2 (0.5)

12. Primary Outcome: Number of Participants With Tolerability Assessment of Scaling
Description: Abnormal shedding of the stratum corneum is measured on a scale 0 to 3. 0 (none) no scaling, 1 (mild) barely perceptible shedding, noticeable only on light scratching or rubbing, 2 (moderate) obvious but not profuse shedding, 3 (severe) heavy scale production. The higher score indicated the worse outcome.
Time Frame: At Week 20
Population: Safety population included all enrolled and randomized participants. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. As per planned efficacy data was separately analyzed and collected for both Metvix cream and Metvix vehicle cream based on 1, 2 and 3 hours group."
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix Cream 160 mg/g (1 Hour Group) | Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g (2 Hour Group) | Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g (3 Hour Group) | Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 11 | 11
Participants
  None | 8 | 8 | 6 | 8 | 7 | 10
  Mild | 1 | 1 | 2 | 1 | 3 | 1
  Moderate | 0 | 0 | 1 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the study drug. Abnormalities presented at Baseline were considered AEs if they reoccurred after resolution or worsen during the AE collection period. Number of participants with AEs were reported.
Time Frame: Up to Week 20
Population: Safety population included all enrolled and randomized participants. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure. As per planned analysis safety data was analyzed and collected for Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group), Metvix Cream 160 mg/g+Metvix Vehicle Cream (2 Hour Group) and Metvix Cream 160 mg/g+Metvix Vehicle Cream (3 Hour Group).
Measure: Number; unit: count of participants
Groups:
- Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 1 hour at Baseline, Weeks 4 and 8. The target area was then exposed to red light LED light source: Aktilite 128 lamp] during 7 to 10 minutes to deliver a total dose of 37 Joules per centimeter square J/cm^2. The total study duration was 20 weeks.
- Metvix Cream 160 mg/g+Metvix Vehicle Cream (2 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 2 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light LED light source: Aktilite 128 lamp] during 7 to 10 minutes to deliver a total dose of 37 Joules per centimeter square J/cm^2. The total study duration was 20 weeks.
Arm/Group | Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group) | Metvix Cream 160 mg/g+Metvix Vehicle Cream (2 Hour Group) | Metvix Cream 160 mg/g+Metvix Vehicle Cream (3 Hour Group)
Number analyzed (Participants) | 11 | 9 | 12
count of participants | 1 | 3 | 8

ADVERSE EVENTS:
Time Frame: From first dose of administration up to Week 20
Description: Safety population included all enrolled and randomized participants. As per planned analysis safety data was analyzed and collected for Metvix Cream 160 mg/g+Metvix Vehicle Cream (1 Hour Group), Metvix Cream 160 mg/g+Metvix Vehicle Cream (2 Hour Group) and Metvix Cream 160 mg/g+Metvix Vehicle Cream (3 Hour Group).
Groups:
- Metvix 160 mg/g Cream+Metvix Vehicle Cream (1 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 1 hour at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix 160 mg/g Cream+Metvix Vehicle Cream (2 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 2 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
- Metvix 160 mg/g Cream+Metvix Vehicle Cream (3 Hour Group): Participants were topically treated with 160 mg/g Metvix cream on one half-face or Metvix vehicle cream on the other half-face for 3 hours at Baseline, Weeks 4 and 8. The target area was then exposed to red light (using a large-field LED light source: Aktilite 128 lamp) during 7 to 10 minutes to deliver a total dose of 37 J/cm^2. The total study duration was 20 weeks.
Arm/Group | Metvix 160 mg/g Cream+Metvix Vehicle Cream (1 Hour Group) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (2 Hour Group) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (3 Hour Group)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/9 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 3/9 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (1 Hour Group) (N=11) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (2 Hour Group) (N=9) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (3 Hour Group) (N=12)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (1 Hour Group) (N=11) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (2 Hour Group) (N=9) | Metvix 160 mg/g Cream+Metvix Vehicle Cream (3 Hour Group) (N=12)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Face Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rash Pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes